CLINICAL TRIAL: NCT00637897
Title: Feasibility of Dose Titrating Paricalcitol (Zemplar) in Women Receiving Taxanes or Ixabepilone for Metastatic Breast Cancer
Brief Title: Paricalcitol and Chemotherapy in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000583652; P30CA012197 (NIH); CCCWFU-74307 (Other: Comprehensive Cancer Center of WFUHS); NCT01055288 (obsolete NCT alias)
Record Dates: First submitted 2008-03-17; First posted 2008-03-18 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; ixabepilone; Paclitaxel; Taxes; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Paricalcitol (Zemplar) (Experimental): Paricalcitol (Zemplar)
  Interventions: Drug: docetaxel; Drug: ixabepilone; Drug: paclitaxel; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: paricalcitol

INTERVENTIONS:
Drug: docetaxel
Drug: ixabepilone
Drug: paclitaxel
Drug: paclitaxel albumin-stabilized nanoparticle formulation
Drug: paricalcitol

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, docetaxel,, paclitaxel, and ixabepilone work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Paricalcitol may help chemotherapy drugs to kill more tumor cells by making tumor cells more sensitive to the drugs.

PURPOSE: This clinical trial is studying the best dose and best way to give paricalcitol and to see how well it works when given together with chemotherapy in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the ability to administer 8 continuous weeks of therapy within the first 3 months of enrollment with paricalcitol when given together with taxane or ixabepilone therapy in women with metastatic breast cancer.
* To estimate the proportion of patients who successfully complete 8 continuous weeks of therapy as well as the proportion of patients who achieve a 'steady-state' dose.

Secondary

* To determine a dose of paricalcitol that can be taken continuously that maintains a normal calcium level when combined with a taxane or ixabepilone.
* To determine if baseline levels of 25-hydroxycholecalciferol and parathyroid hormone (PTH) are associated with time to treatment failure in these patients.
* To determine if PTH levels decline from baseline in patients treated with paricalcitol in combination with taxane or ixabepilone therapy.

OUTLINE: Beginning on day 1, patients receive oral paricalcitol. The dose of paricalcitol is increased every 2 weeks until the serum calcium level is between 9 mg/dL and 11.4 mg/dL. Once this level is reached, the patient continues at that dose for the duration of the study. Patients also receive paclitaxel albumin-stabilized nanoparticle formulation, docetaxel, or paclitaxel once a week or once every 3 weeks or ixabepilone once every 3 weeks. Treatment continues for at least 12 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed invasive breast cancer

  * Metastatic or recurrent disease
  * Patients with bone metastasis only are eligible and evaluable for time to progression
* Candidate for taxane or ixabepilone therapy
* At least one lesion that can be measured in at least one diameter ≥ 2 cm by CT scan
* No symptomatic brain metastases or other symptomatic CNS metastases
* ECOG performance status 0 or 1
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 2.0 g/dL
* Albumin corrected serum calcium < 10.5 mg/dL
* Fertile patients must use effective contraception during and for at least 1 year after study participation
* At least 2 weeks since prior chemotherapy or radiation therapy
* Prior and concurrent taxane or ixabepilone therapy allowed
* Concurrent oral multivitamins allowed (i.e., Centrum or One a Day)
* Concurrent bisphosphonates allowed

Exclusion Criteria

* History of allergy to calcitriol, paricalcitol, or other Vitamin D compounds
* History of drug or alcohol abuse within the past 6 months
* History of other malignancy except inactive nonmelanoma skin cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or other cancer if the patient has been disease-free for 5 or more years
* Serious medical illness that would limit survival to < 3 months
* Active, uncontrolled bacterial, viral or fungal infection
* Poorly controlled diabetes
* Concurrent supplemental calcium
* Concurrent digitalis compounds
* Concurrent chemotherapy
* Concurrent biologic therapy, including trastuzumab and bevacizumab
* Concurrent hormonal agents for breast cancer except luteinizing hormone-releasing hormone agonists

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2011-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Clinical feasibility of therapy administration | Baseline to 8 weeks
  To test the clinical/logistical feasibility of using a titrated dose of the vitamin D analog (paracalcitol or Zemplar) in combination with a taxane or ixabepilone primarily by measuring the proportion of patients who successfully complete 8 continuous weeks of therapy as well as the proportion of patients who achieve a 'steady-state' dose

SECONDARY OUTCOMES:
Dose of paricalcitol that maintains a normal calcium level when given in combination with a taxane or ixabepilone | Baseline to 8 weeks
Correlation of baseline levels of 25-hydroxycholecalciferol and parathyroid hormone with time to treatment failure | Baseline to 8 weeks
  To determine if baseline levels of 25(OH)D and parathyroid hormone are associated with time to treatment failure in patients treated with the combination of paricalcitol and a taxane or ixabepilone
Measurement of effect of combination of paricalcitol and a taxane or ixabepilone on parathyroid hormone levels failure | Baseline to 8 weeks
  To determine if parathyroid hormone levels decline from baseline with the combination of paricalcitol and a taxane or ixabepilone

CONTACTS AND LOCATIONS:
Overall Officials: Julia A. Lawrence, Study Chair — Wake Forest University Health Sciences; Susan A. Melin, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States